CLINICAL TRIAL: NCT03063580
Title: A Phase 1, Single-center, Open-label, 2-period, Single Sequence Drug-drug Interaction Study to Evaluate the Effects of Multiple-dose Rifampicin on the Pharmacokinetics and Pharmacodynamics of Single Dose Sotagliflozin in Healthy Male and Female Subjects
Brief Title: Effect of Rifampicin on the Pharmacokinetics and Pharmacodynamics of Sotagliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INT14936; U1111-1186-2980 (Other: UTN)
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR439954 with or without rifampicin (Experimental): Period 1: single oral dose of 400 mg sotagliflozinon Day 1 morning Period 2: once-daily oral doses of 600 mg rifampicin from Days 1 to 10 and a single oral dose of 400 mg sotagliflozin
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Rifampicin

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablets
  Route of administration: oral
Drug: Rifampicin — Pharmaceutical form: capsules
  Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the effects of rifampicin on the pharmacokinetics (PK) of sotagliflozin and its metabolite in healthy male and female subjects.

Secondary Objectives:

* To assess total 24-hour urinary glucose excretion (UGE) after a dose of sotagliflozin 400 mg, alone and with rifampicin, in healthy male and female subjects.
* To assess the safety and tolerability of single dose sotagliflozin with and without rifampicin in healthy male and female subjects.

DETAILED DESCRIPTION:
The expected duration of the study is approximately 53 days total, including 2-28 days of screening, treatment periods of 6 days and 11 days, 1 day of end of study visit, and at least 7 days of follow-up visit.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, ECG, and laboratory parameters. Total bilirubin out of normal range can be acceptable if total bilirubin should not exceed 1.5 the upper limit with normal conjugated bilirubin values (unless the subject has documented Gilbert syndrome).
* Female subject must use a double contraception method including a highly effective method of birth control, except if she has undergone sterilization at least 3 months earlier or is postmenopausal.
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.

Exclusion criteria:

* Any history or presence of clinically relevant disease at screening, which could interfere with the objectives of the study or the safety of the subject's participation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive β-HCG (human chorionic gonadotropin) blood test if applicable), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion. Any oral contraceptives during the screening period or for at least 15 days prior to inclusion; any injectable contraceptives or hormonal intrauterine devices within 12 months prior to inclusion; or topical controlled delivery contraceptives (patch) for 3 months prior to inclusion.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 96 hours post SAR439954 dosing
Area under the concentration-time curve from 0 to the last quantifiable concentration (AUC0-tlast) | Up to 96 hours post SAR439954 dosing
Area under the concentration-time curve from 0 to infinity (AUC0 ∞) | Up to 96 hours post SAR439954 dosing

SECONDARY OUTCOMES:
Total 24-hour UGE (urinary glucose excretion) | Up to 24 hours after SAR439954 intake

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 250001, Gières, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org